CLINICAL TRIAL: NCT01492543
Title: An Open-label, Single-arm, Multicenter, Phase II Study to Assess the Efficacy and Safety of Aiyi® (Tegafur Gimeracil Oteracil Potassium Capsule) as 2nd Line Treatment in Patients With Advanced Metastatic Breast Cancer
Brief Title: Study of TS-1 as 2nd Line Treatment in Patients With Advanced Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Beijing Chao Yang Hospital (Other); Chinese PLA General Hospital (Other); China-Japan Friendship Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Hebei Tumor Hospital (Other)
Responsible Party: Principal Investigator, Binghe Xu, Deputy Director of Department of Medical Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-014
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: Advanced; Metastatic; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aiyi® (Experimental): Tegafur Gimeracil Oteracil Potassium Capsule
  Interventions: Drug: Tegafur Gimeracil Oteracil Potassium Capsule

INTERVENTIONS:
Drug: Tegafur Gimeracil Oteracil Potassium Capsule — Aiyi® (Tegafur Gimeracil Oteracil Potassium Capsule; T25mg,G7.25mg,O24.5mg*42 capsules/box), manufactured by Jiangsu Hengrui Medicine Co., Ltd.,
  Other Names: TS-1

SUMMARY:
The purpose of this study is to assess the effectiveness and safety profile of Aiyi®(Tegafur Gimeracil Oteracil Potassium Capsule, TS-1) as a second line therapy in Chinese female patients with advanced metastatic breast cancer.

DETAILED DESCRIPTION:
Tegafur Gimeracil Oteracil Potassium Capsule is a novel oral derivative of the 5-fluorouracil(5-FU) prodrug tegafur combined with two modulators. Recent clinical trial has reported the promising effect of Tegafur Gimeracil Oteracil Potassium Capsule in metastatic breast cancer. The innovative drug, S-1, has obtained the approval of treatment of advanced breast cancer in Japan, meanwhile, Generic drug is only approved for the indication of gastric cancer in China mainland by Chinese authority, SFDA, and no Chinese clinical study data of TS-1 in breast cancer so far.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old female.
* ECOG status: 0-2.
* Life expectancy of ≥ 3 months.
* Histologic or cytologic diagnosis of breast cancer.
* Progression after receiving one standard prior chemotherapy regimen for recurrent or metastatic lesion except an endocrine regimen.
* At least one measurable lesion of >=2 cm (>=1 cm on spiral CT scan)according to RECIST (v1.1).
* Adequate organ functions:

  * Hematopoietic: Hemoglobin ≥90g/L, Absolute neutrophil count ≥1.5×10^9/L, Platelet count ≥80×10^9/L.
  * Biochemistry: TBil ≤1.5 times upper limit of normal (ULN), AST and ALT ≤2.5× ULN(≤5x ULN if due to liver metastases), Creatinine ≤1.0×ULN and Creatinine clearance >50 ml/min.
* Women with children potential must have negative pregnancy tests 7 days prior to enrollment and be willing to practice acceptable methods of birth control during the study and 8 weeks after last drug administered.
* Ability to take oral medication .
* Signed informed consent.

Exclusion Criteria:

* Pregnancy or lactation or no effective contraception in fertile patients.
* Prior treatment with 5-FU or drugs of same class(excluding patients that relapsed more than one year after adjuvant therapy).
* Less than 4 weeks since prior investigational agents.
* conditions impacting oral drug taking or absorption (e.g. inability to swallow, gastrointestinal resection, chronic diarrhea, intestinal obstruction).
* Organ invasion with rapid progression(e.g. lesions exceeding half of Liver or Lung).
* CNS or psychiatric disorders.
* Allergic to 5-FU.
* Only with bone metastases and no measurable lesions.
* Clinically significant heart diseases (e.g.congestive heart failure, ventricular arrhythmia, myocardial infarction) before enrollment.
* Serious peptic ulcer disease or digestive disorders.
* Bone marrow (Hemoglobin <90g/dl, ANC <1.5×10^9/L, Platelet count <75×10^9/L).
* Renal function disorder (Creatinine >1.0×ULN).
* Liver function disorder (TBil >1.5×ULN).
* Uncontrolled brain metastases.
* Noncompliance with the study protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 2 years

SECONDARY OUTCOMES:
Clinical response rate | Every six weeks
  Assessed by RECIST v1.1 criteria.
Adverse events | Subjects will be followed from date of enrollment until the date of last visit, anticipated up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (7):
- China (7):
  - Beijing Chao-yang Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Hebei Provincial Tumor Hospital, Shijiazhuang, Hebei
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing